CLINICAL TRIAL: NCT06371079
Title: Safety and Suitability of Implantable Collamer Lens (ICL) Implantation for Correction of Refractive Errors Without the Use of Dispersive Ophthalmic Viscosurgical Devices (OVDs)
Brief Title: Safety and Suitability of ICL for Correction of Refractive Errors Without the Use of Dispersive OVDs
Status: Completed | Type: Observational
Sponsor: Loay Abdulmutalib Almusawi (Other)
Responsible Party: Sponsor-Investigator, Loay Abdulmutalib Almusawi, Ophthalmology Lecturer, University of Basrah
Organization: University of Basrah (Other)
Other Study IDs: NO-OVD-ICL
Record Dates: First submitted 2024-04-06; First posted 2024-04-17 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Refractive Errors; Myopia; Myopic Astigmatism; Hypermetropia
Keywords: refractive errors; myopia; hypermetropia; astigmatism; refractive surgery; ICL; ophthalmic viscosurgical device
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism; Hyperopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Traditional OVD group: In this group of patients, the ICL was implanted utilizing both cohesive and dispersive ophthalmic viscosurgical device.
  Interventions: Device: phakic intraocular lens implantation traditional
- Reduced OVD group: In this group of patients, the ICL was implanted with the use of cohesive OVD only.
  Interventions: Device: phakic intraocular lens implantation reduced OVD

INTERVENTIONS:
Device: phakic intraocular lens implantation traditional — patients with refractive errors undergo surgical implantation of a lens inside the eye (implantable collamer lens or ICL) to correct these refractive errors. The procedure is done with help of use of both cohesive and dispersive OVD
  Other Names: ICL implantation traditional; Intraocular refractive surgery
  Groups: Traditional OVD group
Device: phakic intraocular lens implantation reduced OVD — patients with refractive errors undergo surgical implantation of a lens inside the eye (implantable collamer lens or ICL) to correct these refractive errors. The procedure is done with help of use of only cohesive OVD without using dispersive OVD.
  Other Names: ICL implantation reduced OVD; Intraocular refractive surgery
  Groups: Reduced OVD group

SUMMARY:
The goal of this observational study is to test whether surgeries for lenses designed to be implanted in the eye to correct refractive error can be done without the need for using viscoelastic substances that are used routinely nowadays to make it easier to introduce them inside the human eye and protect the inside of the eye during the operation.

The main question it aims to answer is that is it safe to do the surgery without using them? to answer this question researchers will access recorded data of patients that underwent refractive surgeries in a private clinic since 2017 and compare them as two groups: those who underwent the traditional procedures and those who had it without the use of dispersive viscoelastics in regard to their vision before and after surgery, their ocular pressure and biomicroscopic analysis of the inside of their corneas before and after surgery.

DETAILED DESCRIPTION:
Records of patients that had undergone ICL implantation surgery in Al-Ferdows private eye hospital in Baghdad between 2017 and 2023 were accessed. Two groups of patients were identified, for the first group the ICL was implanted with the use of both dispersive and cohesive OVDs (traditional OVD group) and for the second one a novel method of implantation was used without utilizing dispersive OVD (reduced OVD) group. Both types of surgery were done by the same surgeon and in the same settings. The operative notes of the OVD group were as follows: under topical anesthesia if the ICL is toric, manual corneal marking is done in the sitting position using pendular marker. After loading of the ICL, two-step clear corneal main incision 2.8 mm in width with a bit long track of 1.5-2 mm to enhance its valve action was fashioned. Intracameral injection of dispersive OVD. The ICL was implanted with mouth-to-mouth technique. Anterior chamber reformation with cohesive OVD, then haptics are gently pushed behind the iris using an olive-tipped manipulator, ensuring alignment to proper axis in case of toric ICL, otherwise spherical ICL is placed directly at 180° axis. After that, AC (anterior chamber) wash with irrigation/aspiration is performed then stromal hydration was done to seal the surgical wound. In the reduced OVD group, modification to the traditional method involved omitting the step of dispersive OVD injection and instead utilizing Intracameral injection of 1:1 mixture of 1:1000 adrenaline and 2% lidocaine in an overfilling manner. All other surgical steps are performed in an identical manner.

The study was ethically approved by the institutional review committee at the respective hospital and a similar committee at the college of medicine of university of Basrah according to the local guidelines and protocols. Written informed consent was obtained from each patient before the surgery. The study followed tenets of declaration of Helsinki.

For both groups, records involving preoperative and postoperative assessments such as uncorrected and best corrected visual acuity, refractive error quantification both objectively utilizing an autorefractometer autorefractor Nidek ARK 1 (Nidek Inc, Gamagori, Japan) and subjectively as manifest refraction, clinical slit-lamp examination notes, intraocular pressure with non-contact air puff tonometer Topcon CT-1P (Topcon Inc., Tokyo, Japan), AC depth assessment by Pentacam Scheimpflug (Oculus Optikgeräte GmbH Inc., Wetzlar, Germany), specular microscopy study of corneal endothelial cells (endothelial cell density (ECD), coefficient of variation (CV) and hexagonality) using Topcon SP-1p Specular Microscope (Topcon Corporation, Tokyo, Japan), were accessed and analyzed using the latest software in SPSS. Patients with missing or incomplete data were excluded from the study. Exclusion criteria also included patients with severe ocular surface disease, unstable refraction, glaucoma, cataract, retinal detachment and uveitis. Unpaired t test or Mann-Whitney test was used to compare the two groups according to fulfilled statistical assumptions. Significance was considered at P value less than 0.05.

ELIGIBILITY:
* Inclusion Criteria:
* patients with refractive errors and stable refraction seeking refractive surgery who are fit for phakic IOL (intraocular lens) implantation and having reasonable improvement of visual acuity with refractive correction.

Exclusion Criteria:

* patients with severe ocular surface disease, unstable refraction, glaucoma, cataract, retinal detachment and uveitis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Records of patients that had undergone ICL implantation surgery in Al-Ferdows private eye hospital in Baghdad between 2017 and 2023 were accessed. Two groups of patients were identified, for the first group the ICL was implanted with the use of both dispersive and cohesive OVDs (traditional OVD group) and for the second one, a novel method of implantation was used without utilizing dispersive OVD (reduced OVD) group.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sohaib A Mahmood, FIBMS, Study Chair — Ibn Al-Haithem eye teaching hospital; Loay A Almusawi, FIBMS, Study Director — University of Basrah
Locations (1):
- Al-Ferdows private eye hospital, Baghdad, Iraq

REFERENCES:
- [Background] Peng M, Tang Q, Zhao L, Khan MA, Lin D. Safety of implantable Collamer lens implantation without ophthalmic viscosurgical device: A retrospective cohort study. Medicine (Baltimore). 2020 Jun 12;99(24):e20691. doi: 10.1097/MD.0000000000020691. PMID 32541520
- [Background] Zhang Z, Niu L, Zhao J, Miao H, Chen Z, Shen Y, Chen X, Ye Y, Wang X, Zhou X. Safety of EVO ICL Implantation With an Ophthalmic Viscosurgical Device-Free Technique in the Early 24 h After Surgery. Front Med (Lausanne). 2021 Nov 17;8:764653. doi: 10.3389/fmed.2021.764653. eCollection 2021. PMID 34869472
- [Background] Qin Q, Bao L, He Z, Chen F, Zhu D, Zhang S, Zhang W, Liu Y, Gao R, Xie Z. Pure ICL Implantation: A Novel Ophthalmic Viscosurgical Device-Free Method. J Ophthalmol. 2021 Oct 6;2021:7363267. doi: 10.1155/2021/7363267. eCollection 2021. PMID 34659826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from all patients that had undergone ICL implantation surgery for the correction of refractive errors in Al-Ferdows private eye hospital in Baghdad between 2017 and 2023 were accessed.
Pre-assignment Details: The majority of the enrolled subjects were excluded from the study because most of their data were missing in the records. They cannot be analyzed as per study protocol
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Traditional OVD Group | Reduced OVD Group
Started | 134; 211 Eyes | 314; 446 Eyes
Completed | 46; 78 Eyes | 67; 121 Eyes
Not Completed | 88; 133 Eyes | 247; 325 Eyes
Not completed — Missing data | 88 | 247

BASELINE CHARACTERISTICS:
Population: this involves all participants with complete data
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional OVD Group | Reduced OVD Group | Total
Number analyzed (Participants) | 46 | 67 | 113
Number analyzed (eyes) | 78 | 121 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.04 (7.39) | 29.07 (8.04) | 30.23 (7.90)
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 56 | 79 | 135
  Male | 22 | 42 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 46 | 67 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Iraq | 46 | 67 | 113
Anterior Chamber Depth [Mean (Standard Deviation); unit: Millimeter] — The central depth of the anterior chamber measured in millimeters from the posterior surface of the cornea to the anterior surface of the crystalline lens
  Millimeter | 3.279 (0.299) | 3.308 (0.241) | 3.297 (0.265)
Endothelial Cell Density [Mean (Standard Deviation); unit: cells per square millimeter] — Corneal endothelial cell density as measured using specular microscopy preoperatively
  cells per square millimeter | 2793.75 (310.6) | 2904.56 (307.4) | 2861.47 (312.6)
Corneal endothelial coefficient of variation [Mean (Standard Deviation); unit: unitless] — Defined as the ration of the standard deviation of the corneal endothelial cell size to the mean
  unitless | 29.6 (4.4) | 29.6 (3.9) | 29.6 (4.1)
Corneal endothelial cells hexagonality [Mean (Standard Deviation); unit: percentage] — the percentage of corneal endothelial cells with 6 borders from total number of cells in the analyzed area
  percentage | 58.22 (10.55) | 58.30 (9.77) | 58.27 (10.07)
Central corneal thickness [Mean (Standard Deviation); unit: micrometer] — Central corneal thickness (CCT) as measured using specular microscopy
  micrometer | 493.0 (38.83) | 491.8 (45.60) | 492.3 (42.86)
Intraocular pressure [Mean (Standard Deviation); unit: Millimeters of Mercury] | 15.22 (1.9) | 16.79 (2.7) | 15.98 (2.4)
Unaided visual acuity [Mean (Standard Deviation); unit: LogMAR] — Visual acuity measured using Logmar charts before the procedure without any refractive correction
  LogMAR | 1.170 (0.196) | 1.177 (0.21) | 1.175 (0.20)
Best-corrected Visual acuity [Mean (Standard Deviation); unit: LogMAR] | .33 (.12) | .33 (.11) | .33 (.11)

OUTCOME MEASURES:

1. Primary Outcome: Unaided Visual Acuity After the Procedure
Description: visual acuity (vision of the patient) without use of any glasses measured using LogMar charts. This measure has no specified units
Time Frame: 1-2 years after the surgery
Population: Those are participants with complete data and were considered for final statistical analysis
Measure: Mean (Standard Deviation); unit: LogMar vision
Units Other Than Participants: Eyes
Arm/Group | Traditional OVD Group | Reduced OVD Group
Number analyzed (Participants) | 46 | 67
Number analyzed (Eyes) | 78 | 121
LogMar vision | 0.264 (0.17) | 0.227 (0.12)

2. Secondary Outcome: Intraocular Pressure Postoperatively
Description: intraocular pressure in mmHg as measured by non-contact airpuff tonometer Topcon CT-1P (Topcon Inc., Tokyo, Japan). intraocular pressure is measured in millimeters of mercury
Time Frame: first day, first week and first month after the procedure
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Traditional OVD Group | Reduced OVD Group
Number analyzed (Participants) | 46 | 67
Number analyzed (Eyes) | 78 | 121
mmHg | 17.44 (4.46) | 17.80 (4.58)

3. Secondary Outcome: Specular Microscopy Parameter: Endothelial Cell Density
Description: defined as the number of corneal endothelial cells per square millimeter of area, measured using the automated machine from Topcon SP-1P (Topcon Inc, Tokyo, Japan)
Time Frame: 1-2 years after the surgery
Measure: Mean (Standard Deviation); unit: cells per square millimeter
Units Other Than Participants: Eyes
Arm/Group | Traditional OVD Group | Reduced OVD Group
Number analyzed (Participants) | 46 | 67
Number analyzed (Eyes) | 78 | 121
cells per square millimeter | 2785.4 (417.1) | 2851.0 (305.1)

4. Secondary Outcome: Specular Microscopy Parameter: Endothelial Cells Hexagonality
Description: defined as the percentage of endothelial cells having 6 borders and shaped like a hexagon. this measure reflects the overall health of the endothelial cells and decreased hexagonality below 58-60% indicates corneal enodthelial pleomorphism, also measured using the automated machine from Topcon SP-1P (Topcon Inc, Tokyo, Japan)
Time Frame: 1-2 years after the surgery
Measure: Mean (Standard Deviation); unit: percentage of hexagonal cells
Units Other Than Participants: Eyes
Arm/Group | Traditional OVD Group | Reduced OVD Group
Number analyzed (Participants) | 46 | 67
Number analyzed (Eyes) | 78 | 121
percentage of hexagonal cells | 58.69 (10.43) | 57.93 (9.26)

5. Secondary Outcome: Specular Microscopy Parameter: Coefficient of Variation of Corneal Endothelial Cells
Description: The standard deviation of the mean cell area divided by the mean cell area gives the coefficient of variation, a unitless number that is normally less than 0.30. it reflects the health of endothelial cells and measured using the automated machine from Topcon SP-1P (Topcon Inc, Tokyo, Japan).
Time Frame: 1-2 years after the surgery
Measure: Mean (Standard Deviation); unit: uniteless
Units Other Than Participants: Eyes
Arm/Group | Traditional OVD Group | Reduced OVD Group
Number analyzed (Participants) | 46 | 67
Number analyzed (Eyes) | 78 | 121
uniteless | 27.37 (3.76) | 29.64 (3.85)

6. Other Pre Specified Outcome: Postoperative Complications
Description: such as glaucoma, cataract, persistent uveitis, macular edema, endophthalmitis..etc.
Time Frame: any time post op within the maximum 2 years follow up period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: within one to two years
Description: All-Cause Mortality, and Serious Adverse Events were monitored/assessed for the same population of participants; However, the majority did not complete the study. PIOL implantation surgery carries a very minimal risk of death or life-threatening events and it is performed under topical local anesthesia.
  Still certain ocular adverse events may happen and these may include: glaucoma, cataract, retinal detachment, intraocular inflammation and/or infection, macular edema, corneal damage...etc.
Arm/Group | Traditional OVD Group | Reduced OVD Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/67
Other Adverse Events (participants affected / at risk) | 1/46 | 0/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional OVD Group (N=46) | Reduced OVD Group (N=67)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) — glaucoma defined here as a persistent raise in intra-ocular pressure that would require a medication to lower it back to normal or surgery and it does not resolve on its own (not temporary) with or without glaucomatous optic disc damage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06371079/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT06371079/ICF_001.pdf